CLINICAL TRIAL: NCT06688266
Title: Comparative Effects of Nerve Gliding Exercises and Conventional Grip Strength Exercises on Grip Strength, Range of Motion and Performance of Cricket Batters
Brief Title: Comparative Effects of Nerve Gliding Exercises and Conventional Grip Strength Exercises in Batters.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sehat Medical Complex (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0422
Record Dates: First submitted 2024-10-27; First posted 2024-11-14 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-11

CONDITIONS: Nerve Compression
Keywords: nerve gliding exercises; grip strength; range of motion; hand exercise program
MeSH Terms: conditions — Neuroma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nerve Gilding Exercises (Experimental): Nerve Gilding Exercises
  Interventions: Other: Nerve Gliding Exercises
- Conventional Grip Strength Exercises (Active Comparator): Conventional Grip Strength Exercises
  Interventions: Other: Hand Grip Strength Exercises

INTERVENTIONS:
Other: Nerve Gliding Exercises — This group will receive 25-minute session of nerve gliding exercises per session five days a week for six weeks. It will include: Warm-Up (5 minutes)
  Neural Gliding of the upper quadrant:
  Median nerve glide (5 minutes) Ulnar nerve glide (5 minutes) Radial nerve glide (5 minutes) Cool Down (5 minutes)
  Arms: Nerve Gilding Exercises
Other: Hand Grip Strength Exercises — This group's participants will also receive a 25 -minute session five days per week (for six weeks). Warm-Up (5 minutes) Conventional Grip Strength Exercises (15 Minutes)
  * Tendon gliding sequence of exercises for hand
  * Squeezing a rubber ball or stress ball
  * Dead Hang Cool Down (5 Minutes)
  Arms: Conventional Grip Strength Exercises

SUMMARY:
Cricket is transformed over the years and dynamic of batting has changed. Gone are the days, when batters used to play the game with defensive mindset. Maintaining higher striker rate and arsenal of power hitting is the epitome of stroke play in limited overs cricket.This study will compare the effects of the nerve gliding exercises and conventional grip strength exercises on handgrip strength, range of motion and performance of cricket batters.

It will be a randomized clinical trial where non-probability convenience sampling will be used to recruit participants aged 18 to 35 years from various cricket academies in Lahore.

DETAILED DESCRIPTION:
Cricket is transformed over the years and dynamic of batting has changed. Gone are the days, when batters used to play the game with defensive mindset. Maintaining higher striker rate and arsenal of power hitting is the epitome of stroke play in limited overs cricket. After modernization of the game, several exercises are adapted to enhance the hitting capability of batsmen with conventional grip strength training but the effectiveness of nerve gliding exercises on handgrip strength is not utilized in cricketing population effectively as compared to tennis and squash players, where it improves the efficiency of wrist mobility in efficient stroke play. This study will compare the effects of the nerve gliding exercises and conventional grip strength exercises on handgrip strength, range of motion and performance of cricket batters. It will be a randomized clinical trial where non-probability convenience sampling will be used to recruit participants aged 18 to 35 years from various cricket academies in Lahore.

Participants will be randomized through lottery method and allocated into two groups. Group A (n=20) participants will receive nerve gliding exercises intervention, while Group B (n=20) will receive conventional grip strength exercises intervention. The Adjustable Hand Dynamometer for Grip Strength, Goniometer for Range of motion while Batting Tee Test for performance will be outcome measure tools. Data will be analyzed by SPSS version 26. The normality of the data will be conducted through the Shapiro-Wilk test; for between-group analysis, an independent t-test or Mann-Whitney will be conducted. Similarly, a paired t-test or Wilcoxon Rank test will be conducted for within-group analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 35 years

  * Batsmen
  * Doing net practices more than 4 days per week for at least 3 months.
  * Right hand grip strength (men) 42.9-46.4, Left hand grip strength (men) 42.042.2.

Exclusion Criteria:

* Non-Athletic Population

  * Upper extremity peripheral neuropathies.
  * Tennis/Golfer epicondylitis. Cervical disc herniation.
  * Overuse injuries of the shoulder joint that may affect handgrip strength.
  * Having any neurological or orthopaedical problem related to upper extremity.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-11-30 (Actual); Primary Completion 2025-05-25 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Handgrip Strength Test using Dynamometer | 6 weeks
  A handgrip dynamometer is a device used to measure the strength of a person's hand grip, providing an objective assessment of their hand and forearm muscle strength.
Universal Goniometer | 6 weeks
  A universal goniometer is a medical instrument used to measure the range of motion (ROM) in joints, particularly in the hands and fingers. It consists of a protractor-like device with two arms and a fulcrum, allowing healthcare professionals to quantify the angles formed by joints during movement. Hand goniometer has demonstrated validity as a measure of functional ROM.
Batting Tee Test | 6 weeks
  A batting tee test is a common method used in baseball or softball to assess a player's hitting skills and technique. This test involves the use of a stationary tee, placed at an appropriate height, from which the player hits the ball.

CONTACTS AND LOCATIONS:
Overall Officials: Suleman Ashiq Dr., DPT, MS-SPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amaral CA, Amaral TLM, Monteiro GTR, Vasconcellos MTL, Portela MC. Hand grip strength: Reference values for adults and elderly people of Rio Branco, Acre, Brazil. PLoS One. 2019 Jan 31;14(1):e0211452. doi: 10.1371/journal.pone.0211452. eCollection 2019. PMID 30703162
- [Background] Dodds RM, Syddall HE, Cooper R, Benzeval M, Deary IJ, Dennison EM, Der G, Gale CR, Inskip HM, Jagger C, Kirkwood TB, Lawlor DA, Robinson SM, Starr JM, Steptoe A, Tilling K, Kuh D, Cooper C, Sayer AA. Grip strength across the life course: normative data from twelve British studies. PLoS One. 2014 Dec 4;9(12):e113637. doi: 10.1371/journal.pone.0113637. eCollection 2014. PMID 25474696
- [Background] Incel NA, Ceceli E, Durukan PB, Erdem HR, Yorgancioglu ZR. Grip strength: effect of hand dominance. Singapore Med J. 2002 May;43(5):234-7. PMID 12188074
- See also: Grip strength: effect of hand dominance — https://pubmed.ncbi.nlm.nih.gov/12188074
- See also: Grip strength across the life course: normative data from twelve British studies — https://pubmed.ncbi.nlm.nih.gov/25474696
- See also: Hand grip strength: Reference values for adults and elderly people of Rio Branco, Acre, Brazil — https://pubmed.ncbi.nlm.nih.gov/30703162